CLINICAL TRIAL: NCT03192059
Title: A Phase II Investigation of Pembrolizumab (Keytruda) in Combination With Radiation and an Immune Modulatory Cocktail in Patients With Cervical and Uterine Cancer (PRIMMO Trial)
Brief Title: Study of Pembrolizumab, Radiation and Immune Modulatory Cocktail in Cervical/Uterine Cancer
Acronym: PRIMMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other); Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-001569-97
Record Dates: First submitted 2017-05-29; First posted 2017-06-19 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2018-05

CONDITIONS: Cervical Cancer; Endometrial Cancer; Uterine Cancer
Keywords: Immunotherapy; Radiotherapy; Immune-modulatory cocktail
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Uterine Neoplasms | interventions — pembrolizumab; Radiation; Vitamin D; Aspirin; Lansoprazole; Cyclophosphamide; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): Pembrolizumab, immune modulatory cocktail composed of Vitamin D, Lansoprazole Teva, Cyclophosphamide and Aspirine, radiation and Curcumin
  Interventions: Drug: Pembrolizumab; Radiation: Radiation; Drug: Vitamin D; Drug: Aspirin; Drug: Lansoprazole; Drug: Cyclophosphamide; Dietary Supplement: Curcumin

INTERVENTIONS:
Drug: Pembrolizumab — Efficacy of the combined treatment
Radiation: Radiation — Efficacy of the combined treatment
Drug: Vitamin D — Efficacy of the combined treatment
Drug: Aspirin — Efficacy of the combined treatment
Drug: Lansoprazole — Efficacy of the combined treatment
Drug: Cyclophosphamide — Efficacy of the combined treatment
Dietary Supplement: Curcumin — Efficacy of the combined treatment

SUMMARY:
This is a Phase II study in patients with advanced and/refractory cervical cancer, endometrial carcinoma or uterine sarcoma.

Patients will be treated with an immunomodulatory cocktail (Vitamin D, aspirin, Cyclophosphamide and Lansoprazole), followed by pembrolizumab, combined with radiation. In addition, patients will take Curcumin, a food supplement.

DETAILED DESCRIPTION:
This is a Phase II multi-center, open-label, non-randomized, 3-cohort study in patients with advanced and/or refractory cervical cancer, endometrial carcinoma or uterine sarcoma. Patients will be treated by an immunomodulatory cocktail (consisting of a daily intake of 2000 IU Vitamin D, 325 mg aspirin, 50 mg Cyclophosphamide and 180 or 30 mg Lansoprazole alternating weekly), followed by pembrolizumab administered intravenously at 200 mg in 21-day treatment cycles, combined with radiation (3x 8Gy in 48h-intervals). In addition, patients will take Curcumin, a food supplement on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed endometrial carcinoma, cervical carcinoma or uterine sarcoma, refractory or persistent to chemotherapy or recurrent disease after at least one line of chemotherapy.
* Presence of an index lesion amenable to hypofractionated stereotactic radiotherapy
* At least one lesion outside the radiation field that can be followed by imaging for clinical response according to RECIST and irRC
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion before and after radiotherapy if technically feasible.
* Have a performance status of 0 or 1 or 2 on the ECOG Performance Scale.
* Demonstrate adequate organ function

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2 agent
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks prior to the first dose of trial treatment,
* Known history of active TB (Bacillus Tuberculosis), Human Immunodeficiency Virus (HIV), HTLV or syphilis,non-infectious pneumonitis, has active autoimmune disease.
* Has active central nervous system metastases and/or carcinomatous meningitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate at week 26 | week 26
  Efficacy (objective response rate) at week 26 according to immune related response criteria (irRC)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety according to CTCAE4.0). | up to 30 days post end of study treatment
  The number of unmanageable dose limiting toxicities will be reported for the run-in period and the main trial. This analysis will be performed for both the Full Analysis Set (FAS; evaluable patiënts) and extended FAS (eFAS; all patients included in the trial).
Objective response rate | week 26
  Objective response rate at week 26 according to RECIST criteria
Best OR | week 26
  Best overall response
PFS | up to 156 weeks
  At weeks 26, 52, 75, 104, 130 and 156 the proportion of progression-free patients will be estimated with a 95% confidence interval.
Median PFS | up to 156 weeks
  At weeks 26, 52, 75, 104, 130 and 156 the median PFS will be calculated.
OS | up to 156 weeks
  At weeks 26, 52, 75, 104, 130 and 156 the proportion of patients surviving will be estimated with a 95% confidence interval.
Median OS | up to 156 weeks
  At weeks 26, 52, 75, 104, 130 and 156 the median survival will be calculated.
Quality of life assessment | Quality of life questionnaires will be completed by the patients at baseline, after 3 months of therapy, after 6 months of treatment (end of treatment) and finally 3 months after therapy.
  Quality of life as measured by FACT-Cx questionnaire for the cervical cancer group and by the FACT-G questionnaire for the endometrial carcinoma and uterine sarcoma group. Descriptive statistics of the total score at each visit and the difference with the baseline visit for all other visits will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hannelore Denys, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - University Hospital Antwerp, Antwerp
  - Institut Jules Bordet, Brussels
  - University Hospital Gent, Ghent
  - CMSE Namur, Namur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Jaeghere EA, Hamerlinck H, Tuyaerts S, Lippens L, Van Nuffel AMT, Baiden-Amissah R, Vuylsteke P, Henry S, Trinh XB, van Dam PA, Aspeslagh S, De Caluwe A, Naert E, Lambrechts D, Hendrix A, De Wever O, Van de Vijver KK, Amant F, Vandecasteele K, Verhasselt B, Denys HG. Associations of the gut microbiome with outcomes in cervical and endometrial cancer patients treated with pembrolizumab: Insights from the phase II PRIMMO trial. Gynecol Oncol. 2024 Dec;191:275-286. doi: 10.1016/j.ygyno.2024.10.020. Epub 2024 Nov 7. PMID 39515198
- [Derived] De Jaeghere EA, Tuyaerts S, Van Nuffel AMT, Belmans A, Bogaerts K, Baiden-Amissah R, Lippens L, Vuylsteke P, Henry S, Trinh XB, van Dam PA, Aspeslagh S, De Caluwe A, Naert E, Lambrechts D, Hendrix A, De Wever O, Van de Vijver KK, Amant F, Vandecasteele K, Denys HG. Pembrolizumab, radiotherapy, and an immunomodulatory five-drug cocktail in pretreated patients with persistent, recurrent, or metastatic cervical or endometrial carcinoma: Results of the phase II PRIMMO study. Cancer Immunol Immunother. 2023 Feb;72(2):475-491. doi: 10.1007/s00262-022-03253-x. Epub 2022 Aug 12. PMID 35960332
- [Derived] Tuyaerts S, Van Nuffel AMT, Naert E, Van Dam PA, Vuylsteke P, De Caluwe A, Aspeslagh S, Dirix P, Lippens L, De Jaeghere E, Amant F, Vandecasteele K, Denys H. PRIMMO study protocol: a phase II study combining PD-1 blockade, radiation and immunomodulation to tackle cervical and uterine cancer. BMC Cancer. 2019 May 28;19(1):506. doi: 10.1186/s12885-019-5676-3. PMID 31138229